CLINICAL TRIAL: NCT03366194
Title: The Clinical Efficacy And Safety Of SkinStylus Microneedling System for Ventral Torso Hypertrophic Scars: Clinical Results With 30 Patients
Brief Title: The Clinical Efficacy And Safety Of SkinStylus Microneedling System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esthetic Education LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20172466 2017-002
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Cicatrix, Hypertrophic
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Each participant shall have at least one suitable ventral torso hypertropic scar of sufficient length that it may be easily visualized in two halfs. At the conclusion of the trial all participants shall be provided with a cross over treatment on the non-treated portion of the scar identical to that which was provided within the trial for the purpose of "evening" the ventral torso hypertrophic scar.
Masking Description: 3. The trial shall be blinded and bias minimized in that three (3) physicians who are either dermatologists or plastic surgeons (and not affiliated with the trial or Esthetic Education LLC) shall review the baseline and treatment photographs and score them using the VAS scale (Visual Analogue Scale).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): Each subject shall have a relatively homogenous section of the total scar divided into two relatively equal sides. One side shall be treated with SkinStylus Sterilock System and the other not treated. The side that is chosen for treatment remains constant. The side that is chosen is done so randomly and prior to meeting the subject via a coin flip randomization.
  Interventions: Device: SkinStylus Sterilock System

INTERVENTIONS:
Device: SkinStylus Sterilock System — Microneedling device will be used to treat ventral hypertrophic scars.

SUMMARY:
The purpose of the trial is to provide objective evidence the SkinStylus may be used safely and effectively for the treatment of ventral torso hypertrophic scars.

DETAILED DESCRIPTION:
1. The SkinStylus has been designated as a non-significant risk and therefore will be granted an Investigational Device Exemption (IDE). There are no meaningful changes to the SkinStylus® instructions for use and specifically no new risks will be introduced.
2. Each participant shall have at least one suitable ventral torso hypertropic scar of sufficient length that it may be easily visualized in two halfs. At the conclusion of the trial all participants shall be provided with a cross over treatment on the non-treated portion of the scar identical to that which was provided within the trial for the purpose of "evening" the ventral torso hypertrophic scar. This is entirely voluntary and participants may decline the treatment if they wish.

ELIGIBILITY:
Inclusion Criteria:

1. at least 23 years old
2. shall have at least one suitable ventral torso hypertropic scar of sufficient length that it may be easily visualized in two halfs.
3. The scar(s) must present along a flat surface suitable for application of the SkinStylus® device and consistent medical photography.

Exclusion Criteria:

1. Pregnancy or chance of pregnancy
2. Currently taking Coumadin/Warfarin® or heparin
3. Diagnosis of any type of bleeding disorder
4. Any history of keloid formation
5. Lidocaine, tetracaine, prilocaine, bupivacaine, or benzocaine hypersensitivity
6. Diagnosis of mental disorders requiring inpatient treatment
7. Presence of metal implants around the proposed treatment areas
8. Diagnosis of any undefined wasting disease (Cachexia for example)
9. Diagnosis of an active infection in the treatment area other than mild acne
10. Diagnosis of the presence of tumors or those who are being treated by chemotherapy or radiation therapy
11. Diagnosis of severe cardiovascular and cerebrovascular disease
12. Diagnosis of renal failure

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Stockton, MD, Principal Investigator — Principal Investigator for Esthetic Education LLC
Locations (1):
- Esthetic Education LLC, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SkinStylus Sterilock System Intervention: Each subject shall have a relatively homogenous section of the total scar divided into two relatively equal sides. One side shall be treated with SkinStylus Sterilock System and the other not treated. The side that is chosen for treatment remains constant. The side that is chosen is done so randomly and prior to meeting the subject via a coin flip randomization.
  SkinStylus Sterilock System: Microneedling device will be used to treat ventral hypertrophic scars.
Period: Overall Study
Arm/Group | SkinStylus Sterilock System Intervention
Started | 36
Completed | 34
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 41 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 9
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
Chest vs abdomen [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement Assessed Using the VAS Scar Scoring System
Description: The Visual Analog Scale Scar Scoring System (VAS Scar Scale) is a validated scar assessment scale with a minimum scar improvement value of 0.0 cm on one end of a 10.0 cm long line and 10.0 cm on the other end. The 0.0 cm represents "no change" in the appearance of the scar while 10.0 cm represents "complete resolution" of the scar.
  A panel of 3 expert graders viewed images of the treatment area and the control area before treatment and 90 days after the last treatment. The difference between the measurements taken at baseline and measurements taken two weeks following the end of the treatment of the treatment area was calculated for each participant, for each grader. The difference of all three graders analysis for each subject was averaged. Those participants with a VAS score on the treatment side that met the MCID of an improvement of at least 1.0 cm were identified in the results as "responders". A higher score is a better outcome.
Time Frame: 90 days from date of last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 34
Participants | 22

2. Secondary Outcome: Number of Patients Self-Reporting Improvement Using the Validated Self-Assessed Scar Improvement Scale Satisfaction Survey
Description: The Self-Assessed Scar Improvement Scale is a validated 6-point scale (-1 to 4) describing the patient's opinion regarding the overall improvement of the scar after treatment with "4" constituting the patient believing that the scar had a "75%-99%" improvement, "3" constituting a "50%-75%" improvement, "2" constituting a "25%-50%" improvement, "1" constituting a "1%-25%" improvement, "0" constituting "no change", and "-1" constituting an "exacerbation of the scar's appearance". A higher score means a better outcome.
Time Frame: 90 days from date of last treatment
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Each subject shall have a relatively homogenous section of the total scar divided into two relatively equal sides. One side shall be treated with SkinStylus Sterilock System and the other not treated. The side that is chosen for treatment remains constant. The side that is chosen is done so randomly and prior to meeting the subject via a coin flip randomization.
  SkinStylus Sterilock System: Microneedling device will be used to treat ventral hypertrophic scars.
  Prior to any treatment, each subject shall self-evaluate the appearance of their scar using the validated Self Assessed Scar Improvement Scale.
  90 days after the last treatment, each subject shall self-evaluate the appearance of the treated area of their scar using the validated Self Assessed Scar Improvement Scale.
Arm/Group | Experimental
Number analyzed (Participants) | 34
Participants | 28

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SkinStylus Sterilock System Intervention
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 2/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SkinStylus Sterilock System Intervention (N=34)
Hyperpigmentation transient (Skin and subcutaneous tissue disorders) | 2 (2) — Hyperpigmentation of treatment area that lasts longer than 2 weeks but less than six months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03366194/Prot_SAP_000.pdf